CLINICAL TRIAL: NCT05204329
Title: Safety of Topical Mesenchymal Stromal Cell Secretome for Ocular Surface Disease
Acronym: MSCSecretome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ali R Djalilian, Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0754; 1UG3EY031809-01 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2024-12

CONDITIONS: Mesenchymal Stromal Cells; Cornea; Corneal Defect; Corneal Epithelium Defect
Keywords: Mesenchymal Stromal Cells; Corneal Defect; Corneal Epithelium Defect
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: A longitudinal assessment using a classic dose-escalation study design to evaluate the safety and maximal tolerated dose of topical MSC Secretome eye drops
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose of allogenic MSC drops (Active Comparator): Escalating doses of allogenic MSC eye drops will be assigned at the lowest dose level.
  Interventions: Biological: MSC Secretome Eye Drops
- Medium dose of allogenic MSC drops (Active Comparator): Escalating doses of allogenic MSC eye drops will be assigned at the medium dose level.
  Interventions: Biological: MSC Secretome Eye Drops
- High dose of allogenic MSC drops (Active Comparator): Escalating doses of allogenic MSC eye drops will be assigned at the high dose level.
  Interventions: Biological: MSC Secretome Eye Drops

INTERVENTIONS:
Biological: MSC Secretome Eye Drops — MSC Secretome eye drop will be dispensed.

SUMMARY:
This study is a longitudinal assessment using a classic dose-escalation study design to assess the safety and maximal tolerated dose (MTD) of topical MSC Secretome eye drops. The study will be conducted at Illinois Eye and Ear Infirmary located at University of Illinois at Chicago. The study will use anterior segment Optical Coherence Tomography (OCT)/Scheimpflug Imaging, esthesiometry, and visual analogue scale (VAS) to assess treatment tolerability.

DETAILED DESCRIPTION:
The "Safety of Topical Mesenchymal Stromal Cell Secretome for Ocular Surface Disease" study is designed to evaluate the safety and maximal tolerated dose (MTD) of topical MSC Secretome eye drops in patients with chronic ocular surface disease through a dose-escalation study under a 28-day topical application protocol, and also obtain a preliminary observation on the following:

1. Incidence of treatment emergent adverse events (TEAE) assessed at 28 days following treatment initiation
2. Proportion of patients with improved corneal epithelial barrier at 28 days compared to baseline
3. Final visual acuity, corneal epithelial thickness, corneal stromal haze, corneal sensation, and treatment tolerability

The objective is to determine the dose of MSC Secretome through a first-in-human study through a dose-escalation strategy targeting a toxicity rate of 33% or less.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Chronic corneal epithelial disease with fluorescein staining score ≥ 6 by NEI grading scale
* Reduced corneal sensation (≤ 4 cm measured by Cochet Bonnet esthesiometry) in at least one corneal quadrant
* A stable ocular surface with no objective clinical evidence of significant (> 50%) improvement/worsening of the epithelial disease in the last 30 days
* Epithelial disease refractory to conventional non-surgical treatments (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops; anti-inflammatory therapy)

Exclusion Criteria:

* Any active or suspected ocular infection (bacterial, viral, fungal or protozoal).
* Evidence of corneal ulceration with stromal loss > 10%
* Presence of an epithelial defect ≥1.0 mm in the largest diameter in the affected eye
* Presence of any size epithelial defect that has been persistent for more than 30 days
* Patients unable to discontinue or intermittently remove therapeutic contact lens in the study eye (to apply drops) during the 4-week study period
* History of any ocular surgery (including laser or refractive surgical procedures) in the affected eye within the 3 months prior to study enrollment
* History of chemical injury within the last 6 months prior to study enrollment Known hypersensitivity to one of the components of the study or procedural medications (e.g.,fluorescein)
* History of drug, medication or alcohol abuse or addiction
* Use of any investigational agent within 4 weeks of screening visit
* History of previous enrollment in the MSC Secretome Study at a lower dose
* Participation in another clinical study at the same time as the present study
* Participants who are pregnant at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Epithelial Status Assessment | Day 28
  The primary outcome measure is improved corneal epithelial barrier function at DAY #28assessed by viewing the cornea under slit lamp examination after instillation of sodium fluorescein, assessing the change from baseline in corneal fluorescein staining score. The presence/absence of an epithelial defect on DAY #28 will also be recorded.

SECONDARY OUTCOMES:
Visual Acuity | Baseline, Days 7, 14, 28, 56, 90
  Best-corrected distance visual acuity will be measured using standard ETDRS protocols.
Corneal Epithelial thickness | Baseline, Days 14, 28, 56, 90
  Corneal epithelial thickness measured by anterior segment OCT imaging (Cirrus 6000, Pachymetry, a-scans and b-scans) will assess the treatment effect on thickness on DAY #28 and compared relative to baseline.
Corneal Scarring / Haze | Baseline, Days 14, 28, 56, 90
  Corneal scarring/haze will be assessed via anterior segment OCT imaging (Cirrus 6000; HD cornea, a-scans) to assess the treatment effect on DAY #28 relative to baseline(Images analysis done by Image-J/Metamorph)
Tolerability of MSC secretome drops | Baseline, Days 7, 14, 28, 56, 90
  Drop discomfort will be measured at DAYS #7, #14, and #28 using a visual analogue scale (VAS; range 0 -100), where 0 represents no discomfort and 100 the worst discomfort.
Durability of Corneal Epithelial Status Improvement | Baseline, Days 7, 14, 28, 56, 90
  Durability of the improved corneal epithelial barrier function/integrity will be assessed an outcome measure at DAY #56 and DAY #90. Participants with improved corneal epithelial barrier function/integrity to DAY #28 will be assessed at each subsequent follow-up visits (e.g., DAYS #56, #90) to assess persistence of the healing response.
Time to Improvement of Corneal Epithelial Barrier | Baseline, Days 7, 14, 28, 56, 90
  The time required for an improved epithelial barrier function will be assessed at each visit throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Djalilian, MD, Principal Investigator — University of Illinois at Chicago; Charlotte E Joslin, OD, PhD, Principal Investigator — University of Illinois at Chicago; Elmer Y Tu, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Prockop DJ, Oh JY. Mesenchymal stem/stromal cells (MSCs): role as guardians of inflammation. Mol Ther. 2012 Jan;20(1):14-20. doi: 10.1038/mt.2011.211. Epub 2011 Oct 18. PMID 22008910
- [Background] Mittal SK, Omoto M, Amouzegar A, Sahu A, Rezazadeh A, Katikireddy KR, Shah DI, Sahu SK, Chauhan SK. Restoration of Corneal Transparency by Mesenchymal Stem Cells. Stem Cell Reports. 2016 Oct 11;7(4):583-590. doi: 10.1016/j.stemcr.2016.09.001. Epub 2016 Sep 29. PMID 27693426
- [Background] Wang LT, Ting CH, Yen ML, Liu KJ, Sytwu HK, Wu KK, Yen BL. Human mesenchymal stem cells (MSCs) for treatment towards immune- and inflammation-mediated diseases: review of current clinical trials. J Biomed Sci. 2016 Nov 4;23(1):76. doi: 10.1186/s12929-016-0289-5. PMID 27809910
- [Background] Yun YI, Park SY, Lee HJ, Ko JH, Kim MK, Wee WR, Reger RL, Gregory CA, Choi H, Fulcher SF, Prockop DJ, Oh JY. Comparison of the anti-inflammatory effects of induced pluripotent stem cell-derived and bone marrow-derived mesenchymal stromal cells in a murine model of corneal injury. Cytotherapy. 2017 Jan;19(1):28-35. doi: 10.1016/j.jcyt.2016.10.007. Epub 2016 Nov 10. PMID 27840134
- [Background] Yao L, Li ZR, Su WR, Li YP, Lin ML, Zhang WX, Liu Y, Wan Q, Liang D. Role of mesenchymal stem cells on cornea wound healing induced by acute alkali burn. PLoS One. 2012;7(2):e30842. doi: 10.1371/journal.pone.0030842. Epub 2012 Feb 17. PMID 22363499
- [Background] Roddy GW, Oh JY, Lee RH, Bartosh TJ, Ylostalo J, Coble K, Rosa RH Jr, Prockop DJ. Action at a distance: systemically administered adult stem/progenitor cells (MSCs) reduce inflammatory damage to the cornea without engraftment and primarily by secretion of TNF-alpha stimulated gene/protein 6. Stem Cells. 2011 Oct;29(10):1572-9. doi: 10.1002/stem.708. PMID 21837654
- [Background] Oh JY, Kim MK, Shin MS, Lee HJ, Ko JH, Wee WR, Lee JH. The anti-inflammatory and anti-angiogenic role of mesenchymal stem cells in corneal wound healing following chemical injury. Stem Cells. 2008 Apr;26(4):1047-55. doi: 10.1634/stemcells.2007-0737. Epub 2008 Jan 10. PMID 18192235
- [Background] Ma Y, Xu Y, Xiao Z, Yang W, Zhang C, Song E, Du Y, Li L. Reconstruction of chemically burned rat corneal surface by bone marrow-derived human mesenchymal stem cells. Stem Cells. 2006 Feb;24(2):315-21. doi: 10.1634/stemcells.2005-0046. Epub 2005 Aug 18. PMID 16109757
- [Background] Li F, Zhao SZ. Control of Cross Talk between Angiogenesis and Inflammation by Mesenchymal Stem Cells for the Treatment of Ocular Surface Diseases. Stem Cells Int. 2016;2016:7961816. doi: 10.1155/2016/7961816. Epub 2016 Mar 24. PMID 27110252
- [Background] Cejkova J, Trosan P, Cejka C, Lencova A, Zajicova A, Javorkova E, Kubinova S, Sykova E, Holan V. Suppression of alkali-induced oxidative injury in the cornea by mesenchymal stem cells growing on nanofiber scaffolds and transferred onto the damaged corneal surface. Exp Eye Res. 2013 Nov;116:312-23. doi: 10.1016/j.exer.2013.10.002. Epub 2013 Oct 18. PMID 24145108
- [Background] Eslani M, Putra I, Shen X, Hamouie J, Afsharkhamseh N, Besharat S, Rosenblatt MI, Dana R, Hematti P, Djalilian AR. Corneal Mesenchymal Stromal Cells Are Directly Antiangiogenic via PEDF and sFLT-1. Invest Ophthalmol Vis Sci. 2017 Oct 1;58(12):5507-5517. doi: 10.1167/iovs.17-22680. PMID 29075761
- [Background] Uccelli A, de Rosbo NK. The immunomodulatory function of mesenchymal stem cells: mode of action and pathways. Ann N Y Acad Sci. 2015 Sep;1351:114-26. doi: 10.1111/nyas.12815. Epub 2015 Jul 6. PMID 26152292
- [Background] Coulson-Thomas VJ, Coulson-Thomas YM, Gesteira TF, Kao WW. Extrinsic and Intrinsic Mechanisms by Which Mesenchymal Stem Cells Suppress the Immune System. Ocul Surf. 2016 Apr;14(2):121-34. doi: 10.1016/j.jtos.2015.11.004. Epub 2016 Jan 12. PMID 26804815
- [Background] Maguire G. Stem cell therapy without the cells. Commun Integr Biol. 2013 Nov 1;6(6):e26631. doi: 10.4161/cib.26631. Epub 2013 Sep 27. PMID 24567776
- [Background] Madrigal M, Rao KS, Riordan NH. A review of therapeutic effects of mesenchymal stem cell secretions and induction of secretory modification by different culture methods. J Transl Med. 2014 Oct 11;12:260. doi: 10.1186/s12967-014-0260-8. PMID 25304688
- [Background] Fernandes-Cunha GM, Na KS, Putra I, Lee HJ, Hull S, Cheng YC, Blanco IJ, Eslani M, Djalilian AR, Myung D. Corneal Wound Healing Effects of Mesenchymal Stem Cell Secretome Delivered Within a Viscoelastic Gel Carrier. Stem Cells Transl Med. 2019 May;8(5):478-489. doi: 10.1002/sctm.18-0178. Epub 2019 Jan 15. PMID 30644653
- [Background] Eslani M, Putra I, Shen X, Hamouie J, Tadepalli A, Anwar KN, Kink JA, Ghassemi S, Agnihotri G, Reshetylo S, Mashaghi A, Dana R, Hematti P, Djalilian AR. Cornea-Derived Mesenchymal Stromal Cells Therapeutically Modulate Macrophage Immunophenotype and Angiogenic Function. Stem Cells. 2018 May;36(5):775-784. doi: 10.1002/stem.2781. Epub 2018 Jan 27. PMID 29341332
- [Background] Samaeekia R, Rabiee B, Putra I, Shen X, Park YJ, Hematti P, Eslani M, Djalilian AR. Effect of Human Corneal Mesenchymal Stromal Cell-derived Exosomes on Corneal Epithelial Wound Healing. Invest Ophthalmol Vis Sci. 2018 Oct 1;59(12):5194-5200. doi: 10.1167/iovs.18-24803. PMID 30372747
- [Background] Vizoso FJ, Eiro N, Cid S, Schneider J, Perez-Fernandez R. Mesenchymal Stem Cell Secretome: Toward Cell-Free Therapeutic Strategies in Regenerative Medicine. Int J Mol Sci. 2017 Aug 25;18(9):1852. doi: 10.3390/ijms18091852. PMID 28841158
- [Background] Bara JJ, Richards RG, Alini M, Stoddart MJ. Concise review: Bone marrow-derived mesenchymal stem cells change phenotype following in vitro culture: implications for basic research and the clinic. Stem Cells. 2014 Jul;32(7):1713-23. doi: 10.1002/stem.1649. PMID 24449458
- [Background] Ivy SP, Siu LL, Garrett-Mayer E, Rubinstein L. Approaches to phase 1 clinical trial design focused on safety, efficiency, and selected patient populations: a report from the clinical trial design task force of the national cancer institute investigational drug steering committee. Clin Cancer Res. 2010 Mar 15;16(6):1726-36. doi: 10.1158/1078-0432.CCR-09-1961. Epub 2010 Mar 9. PMID 20215542
- [Background] Cook N, Hansen AR, Siu LL, Abdul Razak AR. Early phase clinical trials to identify optimal dosing and safety. Mol Oncol. 2015 May;9(5):997-1007. doi: 10.1016/j.molonc.2014.07.025. Epub 2014 Aug 14. PMID 25160636
- See also: U.S. Department of Health and Human Services Food and Drug Administration Center for Biologics Evaluation and Research. Considerations for the Design of Early-Phase Clinical Trials of Cellular and Gene Therapy Products. — https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/CellularandGeneTherapy/UCM564952.pdf